CLINICAL TRIAL: NCT00694798
Title: Open Label, Single Arm, Exploratory Phase I Clinical Trial to Evaluate Efficacy and Safety of Mycobacterium w (Mw) in BCG Refractory Superficial Transitional Cell Carcinoma
Brief Title: Study of Mycobacterium w in BCG Refractory Superficial Transitional Cell Carcinoma of Bladder
Acronym: STCC
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cadila Pharnmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-80/8230
Record Dates: First submitted 2008-06-03; First posted 2008-06-11 (Estimated); Last update posted 2012-05-03 (Estimated); Status verified 2012-05

CONDITIONS: Bladder Cancer
Keywords: STCC; Superficial Transitional Cell Carcinoma- BCG refractor
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Mycobacterium w vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mw (Experimental): All enrolled patients to receive Mycobacterium w
  Interventions: Biological: Mycobacterium w

INTERVENTIONS:
Biological: Mycobacterium w — Immunomodulator

SUMMARY:
The primary purpose of this study is to evaluate the response rate of this treatment (Mw) in patients with BCG refractory superficial transitional cell carcinoma. Other objectives include detecting the effect of Mw on Time to Tumor progression and evaluating safety.

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent obtained & signed:

   Ability to understand and the willingness to sign a written informed consent document.
2. Disease characteristics:

   Patients with BCG refractory superficial transitional cell carcinoma, refractory carcinoma in situ, multiple unresected T1 and Ta high grade.

   BCG-refractory STCC is defined as when there is failure to achieve disease-free state at six months after initiation of BCG therapy either as primary or repeat therapy or recurrence of tumor within three months of completion of adequate induction or maintenance therapy or adequate retreatment. .
3. Patient Characteristics:

Age: 18 completed years and above Performance status: ECOG 0-2 Life expectancy: At least 24 weeks Hematopoietic:Hemoglobin ≥ 9.0 g/dL

Co-morbidity

* No patient who has eczema will be allowed to participate in this study.
* Patients who are immuno-compromised will not be enrolled.
* Patients with severe hepatic dysfunctions or with evidence of Cirrhosis will not be enrolled.
* Patients with uncontrolled diabetes mellitus will not be enrolled in the study.

Note: The effects of Investigational product on the developing human fetus at the recommended therapeutic dose are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

Exclusion Criteria:

* Patients who have had cytotoxic chemotherapy or radiotherapy prior to entering the study.
* Intractable urinary tract infection.
* No patient who has eczema should be allowed to participate in this study.
* Patients who are immuno-compromised should not be enrolled.
* Patients with severe hepatic dysfunctions or evidence of Cirrhosis should not be enrolled.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in the study.
* Pregnant women or nursing women are excluded from this study because agents used in the study have potential for teratogenic or abortifacient effects. Because there is known potential risk for adverse events in nursing infants secondary to treatment of the mother with investigational agent, breastfeeding should be discontinued if the mother is treated with investigational product.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmias, or psychiatric illness/social situations that would limit compliance with study requirements.
* Previous splenectomy
* Clinically significant active infection
* Patients with uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Response Rate | 15 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mahesh Desai, MD, Principal Investigator — Muljibhai Patel Urological Hospital; Amillal Bhat, MD, Principal Investigator — S P Medical College & AG of Hospital; Sushil Bhatia, MD, Principal Investigator — Choithram Hospital and Research Centre; Kim Mammen, MD, Principal Investigator — Christian Medical College, Vellore, India; Ketan Rajyaguru, MD, Principal Investigator — Siddhi Vinayak Hospital; Gaurang Gandhi, MD, Principal Investigator — Gandhi Urocare; Kapil Thakkar, MD, Principal Investigator — Excel Hospital; B. R. Shrivastav, MD, Principal Investigator — Cancer Hospital & Research Institute; Anup Kundu, MD, Principal Investigator — IPGMER, S.S.K.M. Hospital; Jitendra Amlani, MD, Principal Investigator — Urocare Hospital; Rasesh Desai, MD, Principal Investigator — Desai Urological and Maternity Hospital; N. K. Mohanty, MD, Principal Investigator — V. M. Medical College and Safdarjang hospital; Shrawan K. Singh, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Ketan Shukla, MD, Principal Investigator — Aarogyam Speciality Hospital; Krishna Moorhty, MD, Principal Investigator — Lourdes hospital; Rajeev Sood, MD, Principal Investigator — Dr. Ram Manohar Lohia Hospital and PGIMER; Purshottam K. Puri, MD, Principal Investigator — Indira Gandhi Medical College, Shimla
Locations (17):
- India (17):
  - Aarogyam Speciality Hospital, Ahmedabad, Gujarat
  - Gandhi Urocare, Ahmedabad, Gujarat
  - Siddhi Vinayak Hospital, Advanced Urology and Orthopedic Centre, Ahmedabad, Gujarat
  - Muljibhai Patel Urological Hospital, Nadiād, Gujarat
  - Urocare Hospital, Rajkot, Gujarat
  - Excel Hospital, Advanced Laproscopy and Urology Centre, Surat, Gujarat
  - Desai Urological & Maternity Hospital, Vadodara, Gujarat
  - Indira Gandhi Medical College, Shimla, Himachal Pradesh
  - Lourdes Hospital, Kochi, Kerala
  - Choithram Hospital and Research Centre, Indore, Madhya Pradesh
  - Cancer Hospital and Research Institute, Gwalior, Madya Pradesh
  - Christian Medical College, Ludhiana, Punjab
  - S.P. Medical College & A. G. of Hospitals, Bikaner, Rajasthan
  - IPGMER, S.S.K.M. Hospital, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education and Research, Chandigarh
  - Dr. Ram Manohar Lohia Hospital & PGIMER, New Delhi
  - V. M. Medical College & Safdarjang Hospital, New Delhi